CLINICAL TRIAL: NCT02039531
Title: THE APPLICATION OF PLASMA RICH IN GROWTH FACTORS FOR KNEE OSTEOARTHRITIS IMPROVES THE QUALITY OF LIFE AND FUNCTIONAL CAPACITY COMPARED WITH CONVENCIONAL TREATMENT WITH VISCOSUPLEMENTATION
Brief Title: Effect Of Plasma Rich In Growth Factors In Knee Osteoarthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Principe de Asturias (Other)
Collaborators: Funds for independent clinical research by the spanish ministry of health (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI 05/2011
Record Dates: First submitted 2013-12-26; First posted 2014-01-17 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-05

CONDITIONS: Knee Osteoarthritis
Keywords: Knee; osteoarthritis; plasma rich in growth factors; platelet rich plasma; hyaluronic acid
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Intercellular Signaling Peptides and Proteins; Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Plasma rich in growth factors (PRGF) (Experimental): Patients in this group will receive one cycle of three intra-articular injections of PRGF every 15 days.
  Procedure for the application of the treatment:
  1. Study Group or PRGF group
  * Blood sample :
    * Taken minimum after 4 hours of fasting and drinking only water in order to maintain low levels of glucose.
    * 20 cc of peripheral blood will be taken by sterile systems with Sodium Citrate buffer to avoid hemolysis.
  * Spinning of the sample:
    * 8 minutes at 1800 rpm .
    * getting the blood fraction containing the PRGF
    * activation of PRGF with 50 ul of 10% CaCl2 per ml of plasma.
    * the application of PRGF should not exceed 90 minutes after the blood sample extraction in order to avoid risk of contamination.
  Interventions: Biological: Plasma rich in growth factors
- Hyaluronic acid (Durolane®) (Active Comparator): Patients in this group will receive a single intra-articular injection at visit 1.
  Interventions: Drug: Hyaluronic Acid

INTERVENTIONS:
Biological: Plasma rich in growth factors
  Arms: Plasma rich in growth factors (PRGF)
Drug: Hyaluronic Acid
  Other Names: Durolane
  Arms: Hyaluronic acid (Durolane®)

SUMMARY:
HYPOTHESIS:

The application of plasma rich in growth factors (PRGF) will improve the quality of life and functional capacity of patients diagnosed with knee osteoarthritis, providing better functional results than conventional treatment with viscosupplementation.

OPERATING ASSUMPTIONS

Following the initial administration of three doses of PRGF interspersed every 15 days, applied via intraarticular, patients will present an improvement in functional test (WOMAC and Lequesne scales) of 15% or more after 6 and 12 months compared to the control group with patients treated with hyaluronic acid.

DETAILED DESCRIPTION:
OBJECTIVES

The overall objective of the study is to assess the effectiveness of the treatment with PRGF in the osteoarthritis of the knee.

Main objective:

- To show more effectiveness after 6 months of the treatment with PRGF, with an improvement in the reference test (WOMAC and Lequesne) of 15 % or more compared to the treatment with hyaluronic acid in patients with osteoarthritis of the knee.

Secondary objectives:

* To assess the effectiveness after 12 months of the treatment with PRGF compared to the treatment with hyaluronic acid.
* To assess the effectiveness after 12 months of the two cycles re-treatment with PRGF (second phase of the study), compared to the effect of a single cycle with PRGF (first phase of the study ).
* Quantifying platelet growth factors blood concentration in patients treated with PRGF and its correlation with the intraarticular effect.

METHODOLOGY.STUDY DESIGN:

First Phase:

A randomized, single-blind, clinical trial will be performed to compare the effectiveness of 2 different treatment strategies (PRGF and hyaluronic acid) in patients with knee osteoarthritis.

Patients will be divided into two homogeneous groups using a randomization procedure by permuted blocks system.

The first group (experimental) will receive the treatment with PRGF; one cycle of three intraarticular doses every 15 days.

The control group, will receive viscosupplementation wih hyaluronic acid of high molecular weight (Durolane®). Its administration is performed in a one cycle of a single intraarticular dose.

Second phase :

An interim analysis of the main objective in the first phase at 6 months will be performed. If the clinical data indicate that the PRGF is more effective than hyaluronic acid and no serious adverse events were described, the investigators will carry out a second phase of extension, exploratory, open label, non randomized, starting-up after 12 months of the finish of the first phase (in order to wash out the effects of the treatment in the first phase). Patients who were treated with hyaluronic acid in the first phase will be offered to be treated with PRGF in two cycles of administration (the first one at the begining and the second one after 6 months) in order to know whether a two-cycles-based-treatment improves the results of a single-cycle-based-treatment.

STUDY VARIABLES

Within the study the investigators will analyze different variables:

Predicting Variables:

* sex
* age
* BMI,
* Grade of chondropathy by classification of Kellgren and Lawrence scale
* laterality
* employment status (Working, unemployed or retired)
* presence of complications.
* quantification of platelet blood concentration in all patients in the study group.

Outcome Variables :

The investigators will use specific tests to evaluate Osteoarthritis of the knee:

* WOMAC scale (Western Ontario and McMaster Universities ).
* Severity index of Lequesne in knee osteoarthritis. Both are tests internationally validated for clinical and functional health assessment in patients with osteoarthritis of the knee. All are translated into spanish and validated by the scientific community for its use in clinical research.
* Visual Analogue Scale (VAS) and SF-363 Health Questionnaire.

The results of the study questionnaires will be measured after 3, 6 and 12 months in both phases.

The WOMAC questionnaire assesses pain intensity in 5 different situations, the joint stiffness in 2 different situations and the functional capacity in 17 everyday situations. Each item is scored from 0 ( "no pain, or without stiffness or no difficulty" ) to 4 ( " Very much " ) . The total score ranges as follows : Pain 0-20 , stiffness 0-8 and Functional Capacity 0-68 .

The severity index of Lequesne for knee osteoarthritis quantifies the severity of disability or severity of osteoarthritis. The pain is measured in 3 items, the maximum distance walked and activities of daily living are measured in 4 situations. Scores ranges from 1-4 (mild inability) to >14 (where the failure is extremely serious).

The SF -36 is a health questionnaire . It is used in medical research. It provides an overview of the state of health of the person. Contains 36 questions addressing different aspects of the daily life of the person.

COLLECTION AND ANALYSIS .

At baseline patients before receiving the first infiltration, regardless of the study group, must complete the tests described earlier. Then, at 3, 6 and 12 months the patients will perform the same tests.

Analysis:

* Description of variables : qualitative variables are summarized by their absolute and relative frequencies. Quantitative variables by its mean and standard deviation, or alternatively, by the median and interquartile range, in case they do not follow normal distribution.
* Comparison of means between the two groups by Student t-test or , alternatively by the U of Mann - Whitney, in case they do not follow normal distribution.
* Qualitative variables will be analyzed using the chi2 test and calculation of relative risk ( RR ) with a 95% of confidence interval.
* Linear regression and correlation between the blood concentration of platelets in the PRGF obtained and injected . These tests will also be conducted to correlate plasma concentrations with these outcome variables.
* Level of statistical significance was set at P < 0.05 .
* The analysis is carried out by intention to treat.

ETHICS

All patients must sign the informed consent before their inclusion. The study was approved by the ethics committee of the Principe de Asturias University Hospital.

The investigators are responsible to ensure the confidentiality of patient's data, and to act according to the Spanish Law of Protection of Personal Data (LO 15/ 1999).

STUDY LIMITATIONS .

Limitations of the study include the lack of control group treated with placebo. In this study a placebo-controlled group is not ethically acceptable, because the patient must undergo invasive procedures with associated risks and discomfort involved. Therefore, in our case we will use as a control group the patients treated with hyaluronic acid, considered as an alternative to surgical treatment of osteoarthritis of the knee .

Another bias that may occur is the loss of patients by different reasons. To prevent this problem, we will contact every month with patients by telephone to remind them the appointments at 3,6 and 12 months.

In the second phase all patients that had completed the first phase in the control group will have the possibility of treatment with two cycles with PRGF. Because it is considered to be very unlikely to remain a residual effect of hyaluronic acid after 12 months of receiving the first infiltration, homogeneity achieved by the randomization in the first phase is expected to be maintained in the second phase. It is considered that 12 months is a relatively short time interval in a longstanding chronic disease such as osteoarthritis of the knee. Just in case, a comparative analysis of the baseline characteristics will be performed and adjusted for differences that may be found. Finally, due to the sample size was estimated to detect a difference between a one cycle treatment with PRGF and hyaluronic acid in the first phase, it is possible that it could be insufficient for comparison in the second phase. Thus, the second phase is considered as exploratory.

ELIGIBILITY:
Inclusion Criteria:

* Age above 55.
* Moderate to severe symptoms according to the WOMAC pain score of more than 6 months of evolution.
* Grade II - III knee osteoarthritis radiographic criteria for the classification of Kellgren and Lawrence.
* BMI Index below 35 which is considered Morbid Obesity according to WHO.
* Absence of treatments for osteoarthritis in the last 6 months.

Exclusion Criteria:

* Patients who have previously received medical treatment through viscosupplementation in the last 6 months.
* Patients who have allergies to some of the components of DUROLANE ® either hyaluronic acid itself or any of its excipients.
* Patients with severe angular changes and joint instability.
* Patients on anticoagulants or antiplatelet treatment that may not temporarily reversed for infiltrations.
* Polyarticular disease
* Infectious Diseases
* Tumor processes on treatment or medical care.
* Immunosuppressive therapy or immunosuppressive processes.
* Inability to understand the health questionnaires and / or adequately complete.

Ages: 55 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2011-08; Primary Completion 2013-02 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Effectiveness after 6 months of treatment with PRGF with an improvement in the reference tests of more than 15% compared to treatment with hyaluronic acid. | 6 months
  Measured by WOMAC and Lequesne reference scales score for osteoarthritis of the knee.

SECONDARY OUTCOMES:
Effectiveness of the treatment with PRGF compared to treatment with hyaluronic acid after 12 months of follow-up. | 12 months
  Measured by the reference tests WOMAC and Lequesne
Effectiveness of the two-cycles-treatment-based with PRGF in the second phase compared to one-cycle-treatment-based in the first phase after 12 months of the second phase | 12 months of follow-up in the second phase
  Measured by the reference scales WOMAC and Lequesne scores
Blood platelet quantification and its correlation with the effect | 12 months (main stage) and 12 months (extension stage)
  To quantify PDGF platelet concentration in patients treated with PRGF and its correlation with the intraarticular effect regarding a single treatment cycle and the two cycles treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Victor Vaquerizo, MD,PhD, Principal Investigator — Hospital Universitario Principe de Asturias
Locations (1):
- Hospital Universitario Principe de Asturias, Alcalá de Henares, Madrid, Spain